CLINICAL TRIAL: NCT06956378
Title: Effects of Emphasizing Instructions on Mental Health Questionnaires
Brief Title: Health Questionnaire Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 6915
Record Dates: First submitted 2025-04-18; First posted 2025-05-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorder (Panic Disorder or GAD); Depression - Major Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instruction Emphasis (Experimental): The second time participants are asked a questionnaire, the study team will emphasize the instructions.
  Interventions: Behavioral: Instruction Emphasis
- Control (No Intervention): Participants will be asked the questionnaire the same way both times

INTERVENTIONS:
Behavioral: Instruction Emphasis — The study team will emphasize the questionnaire instructions when asking the second time.
  Arms: Instruction Emphasis

SUMMARY:
We want to explore if emphasizing certain instructions (i.e. "bothered by") will affect the way participants respond to a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* U.S. resident
* Self-report being treated for or receiving a diagnosis generalized anxiety disorder or major depressive disorder by a licensed provider (e.g., MD, DO, LPCC, LCSW, LMFT) in the past 12 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Day 1
  Study is completed in 1 day. Scale is administered 2 times. Higher scores mean greater depressive symptoms.
Generalized Anxiety Disorder (GAD-7) | Day 1
  Study is completed in 1 day. Scale is administered 2 times. Higher scores mean greater anxiety symptoms.

OTHER OUTCOMES:
Beck's Depression Inventory | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of California - Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No